CLINICAL TRIAL: NCT06268509
Title: Maternal Optimalization on Nutrition for Better Pregnancy Outcomes (MONAS Study)
Brief Title: Nutrition Optimalization Among Pregnant Women to Improve Maternal and Neonatal Outcome in DKI Jakarta
Acronym: MONAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Collaborators: Dinas Kesehatan DKI Jakarta (Unknown); Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Hardya Gustada Hikmahrachim, Principal Investigator, Member of Department of Child Health, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MONAS
Record Dates: First submitted 2024-01-30; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pregnancy Complications; Maternal Death; Preeclampsia; Intrauterine Infection; Pregnancy Hemorrhage; Preterm Birth; Neonatal Death; Low; Birthweight, Extremely (999 Grams or Less); Asphyxia Neonatorum; IUGR
MeSH Terms: conditions — Pregnancy Complications; Maternal Death; Pre-Eclampsia; Premature Birth; Perinatal Death; Birth Weight; Asphyxia Neonatorum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive:
  * Fetomaternal ultrasound examination each trimester by fetomaternal consultants
  * Complete laboratory examination for nutritional panel (complete blood count with reticulocyte profile and iron profile, vitamin D level, zinc level, fatty acid profile, electrophoresis for Thalassemia) as an addition to standard maternal routine laboratory examination
  * Supplements: multivitamin, minerals, vitamin D, fatty acid
  * Intervention regarding any abnormal results of nutritional panel
  * All standard maternal health services according to Indonesian Ministry of Health protocol
  Interventions: Diagnostic Test: Nutritional panel laboratory examination; Dietary Supplement: Pregnancy supplements (other than provided by Ministry of Health); Diagnostic Test: Fetomaternal ultrasound
- Control group (No Intervention): Participants in the control group will receive:
  - All standard maternal health services according to Indonesian Ministry of Health protocol

INTERVENTIONS:
Diagnostic Test: Nutritional panel laboratory examination — As stated in group description
  Arms: Intervention group
Dietary Supplement: Pregnancy supplements (other than provided by Ministry of Health) — As stated in group description
  Arms: Intervention group
Diagnostic Test: Fetomaternal ultrasound — As stated in group description
  Arms: Intervention group

SUMMARY:
The goal of this MONAS Study is to learn about comprehensive monitoring and nutritional intervention among pregnant women in order to improve maternal and neonatal outcomes. The main questions it aims to answer are:

1. Are comprehensive monitoring and nutritional intervention among pregnant women can improve maternal outcomes (maternal death, preterm labour, preeclampsia, intrauterine infection, and bleeding during pregnancy and delivery) compared to standard maternal health services?
2. Are comprehensive monitoring and nutritional intervention among pregnant women can improve neonatal outcomes (neonatal death, low birth weight, intrauterine growth restriction, and neonatal asphyxia) compared to standard maternal health services?

Participants in the intervention group will receive:

* Fetomaternal ultrasound examination each trimester
* Complete laboratory examination for nutritional panel (complete blood count with reticulocyte profile and iron profile, vitamin D level, zinc level, fatty acid profile, electrophoresis for Thalassemia) as an addition to standard maternal routine laboratory examination
* Supplements: multivitamin, minerals, vitamin D, fatty acid
* Intervention regarding any abnormal results of nutritional panel
* All standard maternal health services according to Indonesian Ministry of Health protocol

Participants in the control group will receive:

- All standard maternal health services according to Indonesian Ministry of Health protocol

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy in 1st trimester
* Gestational age less than 10 weeks
* Living in Jakarta greater area
* Agree to participate

Exclusion Criteria:

* Assisted reproductive technology (IVF)
* History of polycystic ovary syndrome
* History of chronic hypertension
* History of diabetes mellitus
* History of preeclampsia in the previous pregnancy
* Had chronic disease: heart disease, autoimmune disease, malignancy, chronic lung disease
* Planning to have delivery outside Jakarta greater area
* Poor obstetric history (miscarriage/ abortion more than 3 times)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Composite of poor maternal outcomes | At anytime between 20 weeks of gestational age until 28 days after delivery
  Number of participants with a combination of maternal death, preterm labour, preeclampsia, intrauterine infection, and bleeding during pregnancy and or after delivery
Composite of poor neonatal outcomes | After delivery of participants (any gestational age) until 28 days of chronological age
  A number of baby born from participants with a combination of neonatal death, low birth weight, intrauterine growth restriction, neonatal asphyxia, and need of admission to intensive care untill 28 daya of age

CONTACTS AND LOCATIONS:
Overall Officials: Rinawati Rohsiswatmo, Prof., M.D., Ph.D., Principal Investigator — Dr Cipto Mangunkusumo Hospital
Locations (1):
- Jakarta Primary Care Health Facility (Puskesmas) under Jakarta Health Office, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided